CLINICAL TRIAL: NCT04216537
Title: Survival Significance and Clinical Characteristics of Molecular Pathology and Genetic Variation in Brain Gliomas
Brief Title: Survival Significance of Molecular Pathology and Genetic Variation in Brain Gliomas
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Zhenyu Zhang, Doctor, The First Affiliated Hospital of Zhengzhou University
Other Study IDs: GiomaMG-1
Record Dates: First submitted 2019-12-31; First posted 2020-01-02 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Glioma; Molecular Sequence Variation; Genetic Change
Keywords: Survival; Subgroup
MeSH Terms: conditions — Glioma | interventions — Genetic Variation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — All participants have signed the informed consent. Fresh frozen tissues of participants are collected immediately after tumor resection and preserved in liquid nitrogen. Whole exome sequencing, RNA sequencing and proteomics are planed to be conducted.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Glioma groups based on molecular pathology or genetic variation — Patients with newly diagnosed glioma that receive tumor resection

SUMMARY:
This study aims to collect clinical, radiological, pathological, molecular and genetic data including detailed clinical parameters, MR and histopathology images, molecular pathology and genetic data. This study seeks to find the prognostic and clinical significance based on molecular and genetic biomarkers/subgroups of gliomas.

DETAILED DESCRIPTION:
Precise classification based on molecular and genetic biomarkers/subgroups for gliomas is challenging. This study aims to collect clinical, radiological, pathological, molecular and genetic data including detailed clinical parameters, MR and histopathology images, molecular pathology (1p/19q co-deletion, MGMT methylation, IDH and TERTp mutations, etc) and genetic data (Whole exome sequencing, RNA sequencing, proteomics, etc). This study seeks to find the prognostic and clinical significance based on molecular and genetic biomarkers/subgroups of gliomas.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have radiologically and histologically confirmed diagnosis of primary glioma
* Life expectancy of greater than 3 months
* Must receive tumor resection
* Must have sufficient fresh frozen tissues for NGS
* Signed informed consent

Exclusion Criteria:

* No gliomas
* No sufficient amount of tumor tissues for detection of molecular pathology
* Patients who are pregnant or breast feeding
* Patients who are suffered from severe systematic malfunctions
* Do not have sufficient fresh frozen tissues for NGS

Ages: 1 Year to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects are all received tumor resection in the First Affiliated Hospital of Zhengzhou University.
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | From enrollment to death of patients. Estimated about 5 years.
  The length of time from enrollment until the time of death (OS, overall survival)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurosurgery, First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Undecided
Undecided